CLINICAL TRIAL: NCT05701228
Title: Casting Light on HOst-cytomegaloviRUs Interaction in Solid Organ Transplantation
Acronym: HORUS
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2022/10
Record Dates: First submitted 2022-12-30; First posted 2023-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Cytomegalovirus Infections; Solid Organ Transplantation
Keywords: immunocompromised hosts; immune response
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood will be collected on day 0, day15, M1, M3, M6, M12 and M24 and at the time of clinical events for CMV requiring additional samples at day 0, M1, M2, M4 of infection (M12 of infection for patients only included at day 0 of infection).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- day 0 of transplantation: This cohort will include 450 patients at the time of transplantation. The following number of participants will be enrolled in the cohort according to strata defined by organ-transplanted type and baseline immune status.
- day 0 of infection: This cohort will include 150 patients at the time of the infection: Approximatively 75 patients will be drawn from the cohort of solid-organ transplant recipients included at day 0 of transplantation. Additional 75 patients developing a CMV infection will be also included.

SUMMARY:
CMV disease remains the most frequent infectious complication post-transplant and it is associated to high morbidity and even mortality. Global efforts from both transplant physicians and researchers in the field is needed to better characterize the host-virus interactions in the transplant setting, with the aim of decreasing the burden of disease and improve the well-being of patients.

"HORUS" (Casting light on HOst-cytomegaloviRUs interaction in Solid organ transplantation) study is a European research project, funded by the European Commission (Horizon Europe) involving 16 partners in seven European countries (France, Spain, Czech Republic, Belgium, Switzerland, Germany and Italy) aiming to better characterize the host-CMV interactions in SOT recipients. The first aim of HORUS study will be to build a European cohort of SOT recipients including clinical characterization and the constitution of a biocollection, which is the aim of HORUS cohort, in order to perform biological, immunological, gene expression, viral kinetics and deep viral genome characterization in the global European HORUS project to improve our understanding of the development of a CMV immune response in the context of immunosuppression.

DETAILED DESCRIPTION:
The overall goal of HORUS study is to improve our understanding of the host-virus relationship of Cytomegalovirus within immunocompromised solid organ transplant recipients in order to propose both knowledge improvement, and clinical immune signatures for decreasing CMV infections/diseases incidence and avoiding the use of toxic antiviral therapy. HORUS' general goal is to enhance our knowledge on risk factors, disease progression and clinical outcomes by analyzing together immune host characteristics, viral characteristics and immunosuppressive drugs. The constitution of two clinical cohorts ("The day 0 of graft cohort" and "the day 0 of infection cohort") will constitute the aim of "HORUS study" with clinical data collection and biocollection which will be used in the global HORUS project to identify immune profiles of patients integrating all the actors involved in viral control, viral and clinical parameters associated with a higher risk of CMV replication and an evolution toward a CMV difficult-to-treat disease.

"HORUS cohorts" is a project of biological samples biobank from solid organ transplant recipients in Hospitals : France (Bordeaux, Toulouse, Paris, Lyon), Spain (Barcelona), Tchequie (Karlova), Italy (Bologna), Switzerland (Lausanne).

Its main objective of this protocol is to collect, prepare, and store

* under CRB conditions (NFS96900) longitudinal biological samples from solid organ transplants (heart, kidney, lung, liver), from day 0 of transplantation and followed for the occurrence of CMV infection.
* Clinical and sociodemographic data associated with this longitudinal biocollection

The secondary objective is to support for the global "HORUS" project aiming at:

* Studying the longitudinal clinical, viral and immunological profile of solid organ transplants after transplantation with or without CMV disease and if CMV disease with or without a "difficult-to-treat" (CMV persistence, relapse, antiviral drug resistance)
* Defining signatures combining virological data, clinical data, donor/recipient data and immune profile of CMV-specific immunity to identify :i) patients at risk of developing CMV infection and ii) at day 0 of infection to identify patient at risk of developing difficult-to-treat CMV infection. The collection of biological samples, associated with the clinico-biological data, to find the global signature constitutes an indispensable step.

ELIGIBILITY:
A cohort 1 of solid-organ transplant recipients at day 0 of transplantation will be included:

* Consecutive patients meeting the following inclusion criteria will be included:

  * Men and women,
  * Age >= 18 years receiving a (living or deceased donor) kidney, lung, liver, and heart allograft,
  * written informed consent obtained from subject,
  * ability to understand and give their written consent,
  * affiliated to health insurance.
* Exclusion criteria would be:

  * D-R- recipients,
  * participant unable or unwilling to comply with study procedures,
  * subjects who are legally detained in an official institution.

A cohort 2 of solid-organ transplant recipients at day 0 of infection:

* Consecutive patients meeting the following inclusion criteria will be included:

  * Men and women,
  * Age >= 18 years receiving a (living or deceased donor) kidney, lung, liver, and heart allograft
  * written informed consent obtained from subject,
  * ability to understand and give their written consent,
  * affiliated to health insurance,
  * post-transplant CMV infection episode.
* Exclusion criteria would be:

  * D-R- recipients,
  * participant unable or unwilling to comply with study procedures,
  * subjects who are legally detained in an official institution.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort 1 will include 450 patients at the time of transplantation:
  Kidney: 6 groups : 50 R+ATG no mTORi, 30 R+ATG mTORi, 50 R+ no ATG no mTORi, 30 R+ no ATG mTORi, 50 D+R- no mTORi, 30 D+R- mTORi Lung: 3 groups of 20 patients R+ ATG,R+ no ATG, D+R- Heart: 3 groups of 30 patients R+ ATG, R+ no ATG, D+R- Liver: 3 groups of 20 patients R+ ATG, R+ no ATG, D+R-
  Cohort 2 will include 150 patients at the time of the infection:
  Approximatively 75 patients are expected to roll-over from the cohort of solid-organ transplant recipients included at day 0 of transplantation (cohort 1).
  Additional 75 patients developing a CMV infection will be also included.
Sampling Method: Non-Probability Sample
Enrollment: 552 (Actual)
Dates: Start 2023-06-26 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Biobank inventory for cohort 1 : day 0 of transplantation | from day of graft (inclusion day) to month 24
  Biobank inventory will be caracterise thanks to : date of collection, date of pre-analytical processing.
Biobank inventory for cohort 1 : day 0 of transplantation | from day of graft (inclusion day) to month 24
  Biobank inventory will be caracterise thanks to : total volume
Biobank inventory for cohort 1 : day 0 of transplantation | from day of graft (inclusion day) to month 24
  Biobank inventory will be caracterise thanks to : number of aliquots for each biological sample: plasma, serum, whole blood, PBMC, biopsies.
Biobank inventory for cohort 1 : day 0 of transplantation | from day of graft (inclusion day) to month 24
  Biobank inventory will be caracterise thanks to : date of extraction
Biobank inventory for cohort 1 : day 0 of transplantation | from day of graft (inclusion day) to month 24
  Biobank inventory will be caracterise thanks to : concentration of DNA and RNA
Biobank inventory for cohort 2 : day 0 of infection | from day of infection (inclusion day) to month 12
  Biobank inventory will be caracterise thanks to : date of collection, date of pre-analytical processing.
Biobank inventory for cohort 2 : day 0 of infection | from day of infection (inclusion day) to month 12
  Biobank inventory will be caracterise thanks to : total volume
Biobank inventory for cohort 2 : day 0 of infection | from day of infection (inclusion day) to month 12
  Biobank inventory will be caracterise thanks to : number of aliquots for each biological sample: plasma, serum, whole blood, PBMC, biopsies,
Biobank inventory for cohort 2 : day 0 of infection | from day of infection (inclusion day) to month 12
  Biobank inventory will be caracterise thanks to : date of extraction,
Biobank inventory for cohort 2 : day 0 of infection | from day of infection (inclusion day) to month 12
  Biobank inventory will be caracterise thanks to : total volume and concentration of DNA and RNA
Biobank inventory for cohort 2 : day 0 of infection | from day of infection (inclusion day) to month 12
  Biobank inventory will be caracterise thanks to : concentration of DNA and RNA
Creation of a Clinical Database | From inclusion day to month 36
  Implementation of a centralized data base with clinical and sociodemographic data from all European clinical sites.

SECONDARY OUTCOMES:
Caracterised the solid organ transplants after transplantation | From inclusion day to month 36
  Assessing the longitudinal clinical profile of solid organ transplants after transplantation with or without a "difficult-to-treat" (CMV persistence)
Caracterised the solid organ transplants after transplantation | From inclusion day to month 36
  Assessing the longitudinal clinical profile of solid organ transplants after transplantation with or without a "difficult-to-treat" (relapse)
Caracterised the solid organ transplants after transplantation | From inclusion day to month 36
  Assessing the longitudinal clinical profile of solid organ transplants after transplantation with or without a "difficult-to-treat" (antiviral drug resistance)
Caracterised the solid organ transplants after transplantation | From inclusion day to month 36
  Assessing the longitudinal viral profile of solid organ transplants after transplantation with or without a "difficult-to-treat" (CMV persistence)
Caracterised the solid organ transplants after transplantation | From inclusion day to month 36
  Assessing the longitudinal viral profile of solid organ transplants after transplantation with or without a "difficult-to-treat" (relapse)
Caracterised the solid organ transplants after transplantation | From inclusion day to month 36
  Assessing the longitudinal viral profile of solid organ transplants after transplantation with or without a "difficult-to-treat" (antiviral drug resistance)
Caracterised the solid organ transplants after transplantation | From inclusion day to month 36
  Assessing the longitudinal immunological profile of solid organ transplants after transplantation with or without a "difficult-to-treat" (CMV persistence)
Caracterised the solid organ transplants after transplantation | From inclusion day to month 36
  Assessing the longitudinal immunological profile of solid organ transplants after transplantation with or without a "difficult-to-treat" (relapse)
Caracterised the solid organ transplants after transplantation | From inclusion day to month 36
  Assessing the longitudinal immunological profile of solid organ transplants after transplantation with or without a "difficult-to-treat" (antiviral drug resistance)
CMV caracterisation | From inclusion day to month 36
  Defining signatures combining virological data profile of CMV-specific immunity to identify patients at risk of developing CMV infection.
CMV caracterisation | From inclusion day to month 36
  Defining signatures combining clinical data profile of CMV-specific immunity to identify patients at risk of developing CMV infection.
CMV caracterisation | From inclusion day to month 36
  Defining signatures combining donor/recipient data profile of CMV-specific immunity to identify patients at risk of developing CMV infection.
CMV caracterisation | From inclusion day to month 36
  Defining signatures combining immune profile of CMV-specific immunity to identify patients at risk of developing CMV infection.
CMV infection caracterisation | From day of infection (inclusion day) to month 36
  Defining signatures combining virological data profile of CMV-specific immunity to identify at day 0 of infection, patient at risk of developing difficult-to-treat CMV infection.
CMV infection caracterisation | From day of infection (inclusion day) to month 36
  Defining signatures combining clinical data profile of CMV-specific immunity to identify at day 0 of infection, patient at risk of developing difficult-to-treat CMV infection.
CMV infection caracterisation | From day of infection (inclusion day) to month 36
  Defining signatures combining donor/recipient data profile of CMV-specific immunity to identify at day 0 of infection, patient at risk of developing difficult-to-treat CMV infection.
CMV infection caracterisation | From day of infection (inclusion day) to month 36
  Defining signatures combining immune profile of CMV-specific immunity to identify at day 0 of infection, patient at risk of developing difficult-to-treat CMV infection.

CONTACTS AND LOCATIONS:
Overall Officials: Laura RICHERT, Pr, Study Chair — Clinical Epidemiology Unit at Bordeaux University Hospital
Locations (7):
- France (7):
  - Hopitel Pellegrin, Bordeaux
  - Hôpital Edouard Hériot, Lyon
  - Hôpital LA PITIE SALPETRIERE, Paris
  - Hôpital Necker, Paris
  - Hôpital Foch, Suresnes
  - Hôpital Rangueil, Toulouse
  - Hôpital Paul Brousse, Villejuif